CLINICAL TRIAL: NCT03090386
Title: Evaluation of Cognitive-Communication Deficits Following Treatment of Primary Brain Tumor Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nadia N. Laack, M.D., PI, Mayo Clinic
Other Study IDs: 16-005834
Record Dates: First submitted 2017-03-10; First posted 2017-03-24 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cognitive Surveys — Complete the Cognitive Communication Survey, standardized cognitive and language assessments, and the Follow-up Cognitive Communication Survey after treatment

SUMMARY:
This study is to evaluate which cognitive-linguistic symptoms are most commonly experienced following brain tumor treatment. Cognitive surveys will be administered after treatment of primary brain tumor cancer.

ELIGIBILITY:
Inclusion Criteria:

* be between18 to 89 years old;
* have undergone at least one cycle of a cancer treatment regimen (e.g., chemotherapy, radiotherapy, surgery)
* have completed at least one cycle of a cancer treatment regimen within five years of enrollment in the study;
* be native speakers of American English;
* have obtained a minimum of a high school education;
* self-report at least one cognitive-linguistic or social-emotional deficit as assessed by the FACT-BR; and
* must demonstrate capacity to sign informed consent based on Informed Consent for Research: A Guide to Assessing a Participant's Understanding tool.

Exclusion Criteria:

* are younger than 18 years old or older than 89 years old;
* have not undergone at least one cycle of a cancer treatment regimen following diagnosis (e.g., chemotherapy, radiotherapy, surgery)
* have not undergone at least one cycle of a cancer treatment regimen in the five year period prior to enrollment;
* are not native speakers of American English;
* have not obtained a minimum of a high school education;
* do not self-report at least one cognitive-linguistic or social-emotional deficit as assessed by the FACT-BR; or
* do not demonstrate the capacity to sign informed consent

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adults diagnosed with a malignant brain tumor either as a primary diagnosis or recurrent
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-25 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Cognitive Communication Survey | 1 day at time of consent
  Survey is completed at time of consent

SECONDARY OUTCOMES:
Cognitive-linguistic Standardized Testing | within 3 months of cognitive communication survey
  Standardized testing will be completed
Follow-up Survey | within 6 months after completion of standardized testing
  Survey will be completed

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials